CLINICAL TRIAL: NCT00384085
Title: All to Target Trial Lantus® (Insulin Glargine) With Stepwise Addition of APIDRA® (Insulin Glulisine) or Lantus With One Injection of Apidra vs a Twice-Daily Premixed Insulin Regimen (Novolog® Mix 70/30) in Adult Subjects With Type 2 Diabetes Failing Dual or Triple Therapy With Oral Agents: a 64-week, Multi-center, Randomized, Parallel, Open-label Clinical Study.
Brief Title: Insulin Glargine "All to Target" Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3515
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Glargine; insulin aspart, insulin aspart protamine drug combination 30:70

ARMS (3):
- Lantus/Apidra-3 (Experimental): Insulin glargine (Lantus) plus up to 3 injections of insulin glulisine (Apidra) added to oral agents.
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine
- Lantus/Apidra-1 (Experimental): Insulin glargine (Lantus) plus up to 1 injection of insulin glulisine (Apidra) added to oral agents.
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Glargine
- Novolog Mix 70/30 (Experimental): Premixed insulin (Novolog® Mix 70/30) added to oral agents.
  Interventions: Drug: Premixed Insulin

INTERVENTIONS:
Drug: Insulin Glulisine — Subcutaneous injection up to 1 injection per day
  Other Names: Apidra
  Arms: Lantus/Apidra-1
Drug: Insulin Glargine — Subcutaneous injection once-a-day
  Other Names: Lantus
  Arms: Lantus/Apidra-1; Lantus/Apidra-3
Drug: Premixed Insulin — Subcutaneous injection twice-a-day.
  Other Names: Novolog Mix 70/30
  Arms: Novolog Mix 70/30
Drug: Insulin Glulisine — Subcutaneous injection up to 3 injections per day.
  Other Names: Apidra
  Arms: Lantus/Apidra-3

SUMMARY:
The primary objectives were:

* To demonstrate the superiority of Lantus plus stepwise addition of mealtime Apidra® (Lantus/Apidra-3) versus twice-daily Premixed insulin based on the proportion of patients achieving target glycemic control (as measured by hemoglobin A1c [HbA1c] <7.0%) at Week 60
* To demonstrate the noninferiority of Lantus plus addition of 1 mealtime Apidra injection (Lantus/Apidra-1) versus twice-daily Premixed insulin based on the reduction from Baseline to Week 60 in HbA1c

ELIGIBILITY:
* Male or female patients
* 30 to 80 years of age
* Body Mass Index <45 kg/m2
* With Type 2 diabetes mellitus for at least 2 years
* With an HbA1c level at screening of >7.5% and >7.0% at randomization
* On stable dual or triple oral therapy for at least 3 months
* Oral agents in 2 or 3 of the following classes: SU or repaglinide, biguanide, or TZD, willing and able to perform self-monitoring of BG
* Females of child-bearing potentially were required to be willing and able to use adequate contraception

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2006-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Polonsky WH, Thompson S, Wei W, Riddle MC, Chaudhari S, Jackson J, Bruno AS. Greater fear of hypoglycaemia with premixed insulin than with basal-bolus insulin glargine and glulisine: patient-reported outcomes from a 60-week randomised study. Diabetes Obes Metab. 2014 Nov;16(11):1121-7. doi: 10.1111/dom.12328. Epub 2014 Jul 12. PMID 24919603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 123 study sites were activated in the United States; 99 sites enrolled and randomized 588 patients from May 2006 to March 2010. 582 patients out of 588 patients were treated. Three sites (which included 26 patients) were found to be non Good Clinical Practices (GCP) compliant.
Pre-assignment Details: Patient were considered enrolled after informed consent were obtained, and randomized after completion of the 4-week run-in phase and assessment of the randomization criteria.
Period: Overall Study
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30
Started | 195 (Randomized) | 196 (Randomized) | 197 (Randomized)
Intent-To-Treat (ITT) | 195 | 196 | 197
Treated (Safety Population) | 194 | 194 | 194
Intent-To-Treat (Excluding nonGCP Sites) | 187 | 186 | 189
Completed | 156 (Based on the entire ITT population) | 150 (Based on the entire ITT population) | 141 (Based on the entire ITT population)
Not Completed | 39 | 46 | 56
Not completed — Adverse Event | 5 | 5 | 4
Not completed — Lack of Efficacy | 0 | 3 | 2
Not completed — No longer Requires Study Treatment | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Lost to Follow-up | 9 | 9 | 10
Not completed — Progressive Disease | 0 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 19 | 29
Not completed — Patient non-compliant | 4 | 4 | 5
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Loss of site personnel | 1 | 0 | 1
Not completed — Sponsor decision | 1 | 2 | 1
Not completed — Patient moved | 1 | 0 | 1
Not completed — Patient required surgery | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30 | Total
Number analyzed (Participants) | 195 | 196 | 197 | 588
Age Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.54) | 53.7 (9.11) | 53.7 (10.65) | 54.1 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 88 | 86 | 252
  Male | 117 | 108 | 111 | 336
Region of Enrollment [Number; unit: participants]
  United States | 195 | 196 | 197 | 588
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 95.2 (19.21) | 97.2 (20.88) | 97.9 (20.49) | 96.8 (20.21)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram/m^2] | 32.7 (5.79) | 33.4 (6.00) | 33.4 (5.62) | 33.1 (5.80)
Duration of diabetes at study entry [Mean (Standard Deviation); unit: years] | 9.4 (6.80) | 9.1 (5.70) | 9.5 (5.87) | 9.3 (6.13)
Age at onset of diabetes [Mean (Standard Deviation); unit: years] | 46.0 (10.74) | 45.1 (9.36) | 44.8 (10.01) | 45.3 (10.05)
Oral antidiabetic treatment combination at study entry [Number; unit: participants]
  sulfonylurea (SU) or meglitinide plus metformin | 97 | 99 | 97 | 293
  SU or meglitinide plus thiazolinedione (TZD) | 9 | 9 | 10 | 28
  TZD plus metformin | 26 | 27 | 27 | 80
  SU or meglitinide plus metformin plus TZD | 63 | 61 | 63 | 187

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) < 7.0% at Week 60 (Lantus/Apidra-3 Versus Novolog Mix 70/30 - Intent To Treat (ITT) Population Without Good Clinical Practices (GCP) Noncompliant Sites)
Description: Responders defined as patients who achieved an HbA1c value <7.0% versus nonresponders. Patients who did not achieve an HbA1c value <7.0% and patients with a missing HbA1c value at Week 60 were considered to be nonresponders.
Time Frame: At week 60
Population: Analysis was performed on Intent-To-Treat population which consisted of all patients who were randomized and for whom there was any post-baseline follow-up information. Patients from nonGCP compliant sites were excluded from this analysis. Additional analysis including those patients were completed to ensure that study results were not compromised.
Measure: Number; unit: percentage of participants
Arm/Group | Lantus/Apidra-3 | Novolog Mix 70/30
Number analyzed (Participants) | 187 | 189
percentage of participants
  HbA1c < 7.0% | 43.3 | 38.6
  HbA1c ≥ 7.0% | 35.3 | 32.3
  Missing data | 21.4 | 29.1
Statistical Analysis 1: Comparison: Lantus/Apidra-3 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0628, Regression, Logistic — The type I error was controlled by performing a 2-tailed comparison at a p=0.0475 level for superiority testing; Adjusted Odds Ratio = 1.56, 95% CI 2-sided [0.97 to 2.52]

2. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 60 (Lantus/Apidra-1 Versus Novolog Mix 70/30)Per Protocol Population
Description: Absolute Change in HbA1c from Baseline to Week 60. If the Week 60 HbA1c evaluation was missing, the patient was counted as having not completed per protocol.
Time Frame: At week 60
Population: Analysis was performed on the Per Protocol (PP) population which included randomized patients who had no major protocol violation and who had HbA1c recorded for both Baseline & Week 60. Patients from non-GCP compliant sites were, by population definition, excluded from this analysis.
Measure: Least Squares Mean (Standard Error); unit: percent HbA1c
Arm/Group | Lantus/Apidra-1 | Novolog Mix 70/30
Number analyzed (Participants) | 138 | 134
percent HbA1c
  baseline HbA1c | 9.30 (0.176) | 9.06 (0.187)
  Absolute change in HbA1c from baseline | -2.30 (0.126) | -1.97 (0.132)
Statistical Analysis 1: Comparison: Lantus/Apidra-1 vs Novolog Mix 70/30; Test type: Non-Inferiority or Equivalence — Noninferiority of Lantus/Apidra-1 would be established if the upper limit of the 2 sided, 99.75% CI for the difference in the mean change from baseline between Lantus/Apidra-1 and Novolog Mix 70/30 was <0.5%; p = 0.0359, Mixed Models Analysis — The type I error was controlled by performing a 2-tailed comparison at a p=0.0025 level for noninferiority testing; Adjusted Mean of difference = -0.34, 95% CI 2-sided [-0.82 to 0.15]

3. Primary Outcome: Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) < 7.0% at Week 60 (Lantus/Apidra-3 Versus Novolog Mix 70/30 - ITT Population With All Sites) (Sensitivity Analysis)
Description: as for outcome 1
Time Frame: At week 60
Population: Analysis was performed on the Intent To Treat (ITT) population which consisted of all patients who were randomized, and for whom there was any post-baseline follow-up information. Patients from non-GCP compliant sites were included in this analysis. This analysis was performed to ensure that study results were not compromised.
Measure: Number; unit: percentage of participants
Arm/Group | Lantus/Apidra-3 | Novolog Mix 70/30
Number analyzed (Participants) | 195 | 197
percentage of participants
  HbA1c < 7.0% | 44.1 | 38.1
  HbA1c ≥ 7.0% | 34.4 | 32.0
  Missing data | 21.5 | 29.9
Statistical Analysis 1: Comparison: Lantus/Apidra-3 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0313, Regression, Logistic — The type I error was controlled by performing a 2-tailed comparison at a p=0.0475 level for superiority testing; Adjusted Odds Ratio = 1.66, 95% CI 2-sided [1.04 to 2.64]

4. Secondary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 60 (Lantus/Apidra-3 Versus Novolog Mix 70/30)
Description: Absolute Change in HbA1c from Baseline to Week 60.
Time Frame: From baseline to week 60
Population: Analysis was performed on the modified ITT (mITT) population which consisted of all patients who were randomized, and for whom there was a baseline observation and at least 1 postbaseline (on therapy) observation for HbA1c. Patients from non-GCP compliant sites (8 from Lantus/Apidra-3 & 7 from Novolog Mix arms) were excluded from this analysis.
Measure: Least Squares Mean (Standard Error); unit: percent HbA1c
Arm/Group | Lantus/Apidra-3 | Novolog Mix 70/30
Number analyzed (Participants) | 144 | 134
percent HbA1c | -2.45 (0.134) | -2.13 (0.142)
Statistical Analysis 1: Comparison: Lantus/Apidra-3 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0565, ANCOVA; Adjusted Mean of difference = -0.31, 95% CI 2-sided [-0.63 to 0.01]

5. Secondary Outcome: Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) <7.0% at Week 60 (Lantus/Apidra-1 Versus Novolog Mix 70/30)
Description: Patients who achieved an HbA1c value <7.0% were defined as responders. Patients who did not achieve HbA1c values <7.0% and patients with missing HbA1c values were considered nonresponders.
Time Frame: At week 60
Population: Analysis was performed on the modified intent-to-treat population which consisted of all patients who were randomized & for whom there was a baseline observation & at least 1 postbaseline (on therapy) observation for HbA1c. Patients from non-GCP compliant sites (9 for Lantus/Apidra-1 & 7 for Novolog Mix arms) were excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lantus/Apidra-1 | Novolog Mix 70/30
Number analyzed (Participants) | 180 | 185
percentage of participants | 51.1 | 39.5
Statistical Analysis 1: Comparison: Lantus/Apidra-1 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0140, Regression, Logistic; Adjusted Odds Ratio = 1.79, 95% CI 2-sided [1.12 to 2.85]

6. Secondary Outcome: Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) <7.0% at Week 60 Without a Severe Hypoglycemic Event or a Symptomatic Hypoglycemic Event With an Self Monitoring Blood Glucose (SMBG) <50 mg/dl
Description: Severe hypoglycemia was defined as an event with clinical symptoms that are considered to result from hypoglycemia in which the patient required assistance of another person and one of the following: the event was associated with a measured blood glucose level below 36 mg/dL or the event was associated with prompt recovery after oral carbohydrate, iv glucose, or glucagon administration.
  A symptomatic hypoglycemic event was defined as a hypoglycemic episode with an associated SMBG value of <50 mg/dL with reported symptoms.
Time Frame: At week 60
Population: Analysis was performed on the mITT population. Patients from non-GCP compliant sites (8 from Lantus/Apidra-3, 9 from Lantus/Apidra-1 & 7 from Novolog Mix arms) were excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30
Number analyzed (Participants) | 183 | 180 | 185
percentage of participants
  HbA1c < 7.0% | 23.0 | 25.0 | 14.1
  HbA1c ≥ 7.0% | 55.7 | 52.2 | 58.4
  Missing data | 21.3 | 22.8 | 27.6
Statistical Analysis 1: Comparison: Lantus/Apidra-3 vs Lantus/Apidra-1; Test type: Superiority or Other; p = 0.9268, Regression, Logistic; Adjusted Odds Ratio = 1.02, 95% CI 2-sided [0.61 to 1.71]
Statistical Analysis 2: Comparison: Lantus/Apidra-3 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0107, Regression, Logistic; Adjusted Odds Ratio = 2.11, 95% CI 2-sided [1.19 to 3.73]
Statistical Analysis 3: Comparison: Lantus/Apidra-1 vs Novolog Mix 70/30; Test type: Superiority or Other; p = 0.0121, Regression, Logistic; Adjusted Odds Ratio = 2.06, 95% CI 2-sided [1.17 to 3.61]

7. Secondary Outcome: Adjusted Incidence Rate of Hypoglycemia
Description: Adjusted incidence rate of hypoglycemia: estimated percent of patients having at least 1 event of a given type of hypoglycemia.
  A severe Hypoglycemic Event (HE) is one where patient requires assistance. It is confirmed either by a prompt response to certain countermeasures or by a blood Glucose (BG) <36 mg/dL during or soon after the event.
  A serious HE is one where the patient has loss of consciousness, coma, seizure, or convulsion.
  Nocturnal = events occurring between 00:00 & 06:00 based on a 24-hour clock.
  An event is included if the HE start date is within the treatment period.
Time Frame: Week 60
Population: The analysis was performed on the exposed population (i.e. safety population) regardless of enrollment in a non-GCP compliant site.
Measure: Mean (Standard Error); unit: estimated percentage per patient
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30
Number analyzed (Participants) | 194 | 194 | 194
estimated percentage per patient
  Self-Monitored Blood Glucose (SMBG) < 70 mg/dl | 74.40 (3.83) | 74.78 (3.80) | 83.15 (3.11)
  SMBG< 70 mg/dl with symptoms | 60.14 (4.24) | 62.50 (4.18) | 71.98 (3.76)
  SMBG< 70 mg/dl, nocturnal | 46.30 (4.28) | 40.31 (4.18) | 42.53 (4.19)
  SMBG< 70 mg/dl with symptoms, nocturnal | 37.03 (4.10) | 33.55 (3.98) | 35.68 (4.03)
  SMBG< 50 mg/dl | 39.77 (4.27) | 39.55 (4.25) | 53.14 (4.33)
  SMBG< 50 mg/dl with symptoms | 31.51 (3.95) | 32.56 (4.00) | 45.92 (4.30)
  SMBG< 50 mg/dl, nocturnal | 12.05 (2.88) | 11.29 (2.78) | 12.58 (2.96)
  SMBG< 50 mg/dl with symptoms, nocturnal | 6.93 (2.28) | 7.49 (2.43) | 8.88 (2.76)
  SMBG< 36 mg/dl | 10.89 (2.23) | 8.63 (2.02) | 14.32 (2.52)
  Severe hypoglycemias | 10.10 (2.17) | 7.19 (1.85) | 8.23 (1.97)
  Serious hypoglycemias | 0.41 (0.43) | 0.00 (0.00) | 2.29 (1.12)

8. Secondary Outcome: Adjusted Hypoglycemic Event Rates (Event/Patient-year)
Description: Adjusted Hypoglycemic event rate: Total # of events for a given type of hypoglycemia divided by the total exposure to study drug (patient-years). Rates are estimated from a general linear model adjusted for baseline BMI and oral agent combination of antidiabetic medications on which the patient entered the study.
  An event is included if the hypoglycemic event start date is within the treatment period (i.e., from the Randomization date to & including 1 day after the date of last dose of study drug).
Time Frame: Week 60
Population: as for outcome 7
Measure: Mean (Standard Error); unit: event per patient year
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30
Number analyzed (Participants) | 194 | 194 | 194
event per patient year
  Self-Monitored Blood Glucose (SMBG) < 70 mg/dl | 14.50 (1.72) | 12.85 (1.50) | 20.42 (2.38)
  SMBG< 70 mg/dl with symptoms | 7.23 (0.99) | 7.11 (0.99) | 12.23 (1.68)
  SMBG< 70 mg/dl, nocturnal | 1.90 (0.32) | 1.84 (0.31) | 1.68 (0.29)
  SMBG< 70 mg/dl with symptoms, nocturnal | 1.16 (0.21) | 1.10 (0.21) | 1.16 (0.23)
  SMBG< 50 mg/dl | 1.38 (0.21) | 1.17 (0.19) | 2.42 (0.36)
  SMBG< 50 mg/dl with symptoms | 0.89 (0.15) | 0.83 (0.15) | 1.91 (0.31)
  SMBG< 50 mg/dl, nocturnal | 0.20 (0.06) | 0.18 (0.06) | 0.27 (0.09)
  SMBG< 50 mg/dl with symptoms, nocturnal | 0.10 (0.04) | 0.09 (0.04) | 0.18 (0.07)
  SMBG< 36 mg/dl | 0.15 (0.03) | 0.10 (0.03) | 0.23 (0.05)
  Severe hypoglycemias | 0.17 (0.05) | 0.10 (0.03) | 0.17 (0.05)
  Serious hypoglycemias | NA (NA) — Model did not fit data adequately to produce reliable results | NA (NA) — Model did not fit data adequately to produce reliable results | NA (NA) — Model did not fit data adequately to produce reliable results

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent Form up to the last visit were collected.
Description: The analysis was performed on the exposed population (i.e. safety population) and included all AE that developed/worsened during the 'on-treatment period' (i.e. from randomization up to 24 hours after treatment discontinuation or final follow-up visit, whichever came first) regardless of enrollment in a non-GCP compliant site.
Arm/Group | Lantus/Apidra-3 | Lantus/Apidra-1 | Novolog Mix 70/30
Serious Adverse Events (participants affected / at risk) | 22/194 | 23/194 | 21/194
Other Adverse Events (participants affected / at risk) | 140/194 | 150/194 | 152/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lantus/Apidra-3 (N=194) | Lantus/Apidra-1 (N=194) | Novolog Mix 70/30 (N=194)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 3 | 2
Angina unstable (Cardiac disorders) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Faecalith (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Diabetic coma (Nervous system disorders) | 0 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lantus/Apidra-3 (N=194) | Lantus/Apidra-1 (N=194) | Novolog Mix 70/30 (N=194)
Any gastrointestinal disorders (Gastrointestinal disorders) | 33 | 32 | 30
Diarrhoea (Gastrointestinal disorders) | 10 | 10 | 5
Any general disorders and administration site conditions (General disorders) | 21 | 28 | 25
Oedema peripheral (General disorders) | 14 | 11 | 10
Any infections and infestations (Infections and infestations) | 66 | 82 | 90
Bronchitis (Infections and infestations) | 8 | 12 | 12
Nasopharyngitis (Infections and infestations) | 15 | 17 | 8
Sinusitis (Infections and infestations) | 6 | 19 | 16
Upper respiratory tract infection (Infections and infestations) | 18 | 20 | 25
Any musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 45 | 44 | 40
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 12 | 10
Any nervous system disorders (Nervous system disorders) | 39 | 29 | 27
Headache (Nervous system disorders) | 6 | 10 | 5
Any respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.